CLINICAL TRIAL: NCT05974969
Title: A Randomized, Double-Blind, Comparative Clinical Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of Single Intravenous Infusion of BCD-264 and Darzalex® in Healthy Volunteers
Brief Title: A Study to Assess the PK, PD, Safety and Immunogenicity of Single IV Infusion of BCD-264 and Darzalex in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BCD-264-1
Record Dates: First submitted 2023-06-28; First posted 2023-08-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-264 (Experimental): INN: daratumumab, single IV infusion at a dose of 8 mg/kg.
  Interventions: Drug: BCD-264
- Darzalex (Active Comparator): INN: daratumumab, single IV infusion at a dose of 8 mg/kg.
  Interventions: Drug: Darzalex

INTERVENTIONS:
Drug: BCD-264 — a single intravenous infusion of BCD-264
  Arms: BCD-264
Drug: Darzalex — a single intravenous infusion of Darzalex
  Arms: Darzalex

SUMMARY:
The goal of this clinical study is to establish the comparability of the pharmacokinetics and similarity of the safety, immunogenicity and pharmacodynamic profiles of BCD-264 and Darzalex following a single intravenous infusion in healthy subjects.

DETAILED DESCRIPTION:
In this clinical study, each subject will receive a single intravenous infusion of BCD-264 or Darzalex, depending on the group the subject will be randomized to. The drugs are administered at the study site at a dose of 8 mg/kg.

The subjects will be followed up and blood samples collected for pharmacokinetics, pharmacodynamics, immunogenicity and safety studies up to and including 71 study days after the administration of IP.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Men aged 18-45 years inclusive at the time of signing the Informed Consent Form.
3. Body mass index (BMI) in the range of 18.5-30.0 kg/m2.
4. The confirmed "healthy" status based on the conventional clinical and laboratory assessments and investigations obtained as screening.
5. Hemodynamic parameters within the normal range: systolic blood pressure (SBP) in the range of 100-130 mmHg, diastolic (DBP) in the range of 60-90 mmHg, wrist pulse rate 60-90 bpm, obtained at screening.
6. The ability of the subject to follow the Protocol procedures, according to the Investigator.
7. No history of alcoholism abuse or drug addiction and negative test results for alcohol, psychotropic and narcotic substances, psychoactive drugs at screening and before IP infusion.
8. The willingness of subjects, starting from the moment of signing the informed consent form, during the study and for 3 months after the IP administration, to use condoms during any sexual contact by penetration with persons of any sex, including pregnant women. This requirement does not apply to participants who underwent surgical sterilization (bilateral orchiectomy).
9. Willingness to refuse to donate sperm and to conceive a child starting from signing the informed consent form, during the study and for 3 months after the IP administration.
10. Willingness to refrain from drinking alcohol a day (24 hours) before the IP administration and for 96 hours after the administration, and then a day before each scheduled visit.
11. Willingness to refrain from smoking within 2 hours before the IP administration and then 2 hours before each measurement of blood pressure (BP), pulse rate at the wrist, respiratory rate, blood sampling, ECG.
12. Willingness to refrain from vaccination with live attenuated vaccines (intranasal influenza, measles, mumps, rubella, polio, BCG, yellow fever, chickenpox, and typhoid TY21a vaccines) during the main study period.
13. Willingness to refrain from taking any medications, including over-the-counter drugs, vitamins and food supplements, with the exception of drugs prescribed by the investigator for the treatment of AEs, throughout the study.
14. Willingness to refrain from donating blood and plasma for 6 months after the IP administration.

Exclusion Criteria:

1. Mental illness or other conditions that may affect the subject's ability to comply with the Study Protocol.
2. Any surgery performed less than 30 days before the screening.
3. Impossibility to insert a venous catheter for blood sampling (for example, due to skin disease at venipuncture sites).
4. History of severe hypersensitivity reactions (anaphylaxis or multiple drug allergy).
5. Known allergy or intolerance to monoclonal antibody products (murine, chimeric, humanized, and fully human) or any other components of the IP.
6. Administration and use of the following drugs:

   * Regular oral or parenteral administration of any medicinal products, including over-the-counter drugs, vitamins, and dietary supplements, within less than 14 calendar days prior to estimated date of randomization;
   * A history of receiving daratumumab and/or other anti-CD38 monoclonal antibodies.
   * Taking medications, including over-the-counter drugs that have a pronounced effect on hemodynamics and liver function (barbiturates, omeprazole, cimetidine, etc.), within less than 30 days before the estimated date of randomization.
   * Taking drugs that affect the immune status (cytokines and their inducers, glucocorticoids, etc.) within less than 60 days before the estimated date of randomization.
   * Systemic use of antibacterial, antimycotic, antiviral or antiprotozoal drugs within less than 60 days before the estimated date of randomization.
7. Positive results of screening tests for HIV, hepatitis B and C viruses.
8. Positive result of indirect antiglobulin test (indirect Coombs test) at screening.
9. Conventional laboratory parameters or investigations out of the reference ranges accepted at the study sites.
10. Chronic diseases of the cardiovascular, bronchopulmonary, and neuroendocrine systems, as well as diseases of the gastrointestinal tract, kidneys, and blood.
11. Acute infectious diseases less than 4 weeks before the estimated date of randomization, as well as chronic and other diseases that, in the Investigator's opinion, may affect the PK parameters and safety of the IP.
12. Smoking over 10 cigarettes a day.
13. Consumption of more than 10 units of alcohol a week (1 unit of alcohol is equivalent to ½ L of beer, 200 mL of wine or 50 mL of spirits) or a history of alcoholism, drug addiction, or drug abuse.
14. Donation of ≥450 mL of blood or plasma within 60 calendar days prior to the expected date of randomization;
15. Participation in any clinical studies of medicinal products at the time of signing the informed consent or less than 30 calendar days before the expected date of randomization, if the subject received the medicinal product during the clinical study.
16. Previous participation in the same study if the subject was randomized and received the IP during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to infinity (AUC0-∞) | Up to Day 71

SECONDARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to the last measurable concentration (AUC0-t) | Up to Day 71
Maximum observed drug concentration (Cmax) | Up to Day 71
Time from administration to maximum observed concentration of the drug (Тmax) | Up to Day 71
Elimination half-life (Т½) | Up to Day 71
Elimination rate constant (Кel) | Up to Day 71
Total clearance (Cl) | Up to Day 71
Volume of distribution (Vd) | Up to Day 71
Maximum effect (Emax) | Up to Day 71
  Pharmacodynamics will be evaluated based on the absolute count and percentage of CD38+ cells in peripheral blood (T cells, B cells, NK cells, plasmablasts and plasma cells)
Time to maximum effect (TEmax) | Up to Day 71
  Pharmacodynamics will be evaluated based on the absolute count and percentage of CD38+ cells in peripheral blood (T cells, B cells, NK cells, plasmablasts and plasma cells)
Incidence and characteristics of adverse events | Up to Day 71
Proportion of subjects with BAbs/NAbs | Up to Day 71
Time until the BAb/NAb development | Up to Day 71

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Institute of the Human Brain n. a. N.P. Bekhtereva Russian Academy of Sciences, Saint Petersburg
  - Smorodintsev Research Institute of Influenza, Saint Petersburg
  - X7 Clinical Research, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No